CLINICAL TRIAL: NCT02832869
Title: Impact of Reinforced Education by Wechat and Short Message Service on the Quality of Bowel Preparation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director, Head of Department of Gastroenterology, Principal Investigator, Clinical Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Wechat-01
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Bowel Preparation Scale; Adenoma Detection Rate
Keywords: Polyp detection rate; Adenoma detection rate; Boston Bowel Preparation Scale

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- short message service (Experimental): The patients will receive standard written instructions on preparing for a colonoscopy plus intervention such as short message system based re-education by one investigator on the day before colonoscopy.
  Interventions: Other: short message service based re-education
- Wechat (Experimental): The patients will receive standard written instructions on preparing for a colonoscopy plus intervention such as Wechat based re-education by one investigator on the day before colonoscopy.
  Interventions: Other: Wechat based re-education
- Standard preparation instructions (No Intervention): The control arm will receive written instruction on preparing for a colonoscopy per standard of care

INTERVENTIONS:
Other: short message service based re-education — The patients will receive standard written instructions on preparing for a colonoscopy plus intervention such as short message system based re-education by one investigator on the day before colonoscopy.
  Arms: short message service
Other: Wechat based re-education — The patients will receive standard written instructions on preparing for a colonoscopy plus intervention such as Wechat based re-education by one investigator on the day before colonoscopy.
  Arms: Wechat

SUMMARY:
High quality bowel preparation is essential for successful colonoscopy. This study aimed to assess the impact of reinforced education by Wechat or short message service (SMS) on the quality of bowel preparation. This prospective, endoscopist-blinded, randomized, controlled study was conducted. Reinforced education groups received additional education via reminders by Wechat or SMS 2 days before colonoscopy. The primary outcome was the quality of the bowel preparation according to the Boston Bowel Preparation Scale (BBPS). The secondary outcomes included polyp detection rate (PDR), adenoma detection rate (ADR), tolerance, and subjective feelings of patients.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-80 years
* can access to Wechat themselves or through close family members living in the same household

Exclusion Criteria:

* inpatients
* pregnancy
* breast feeding
* history of colorectal surgery
* patients allergic to PEG-ELS based laxatives

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Quality of bowel preparation using Boston Bowel Preparation Scale | 1 day
  The primary outcomes will be the endoscopist's assessment of the quality of preparation using Boston Bowel Preparation Scale

SECONDARY OUTCOMES:
polyp detection rate | 1 day
  The number of polyp prescribed by endoscopist
Patient compliance using a pre-procedure questionnaire | 1 day
  Patient compliance with preparation instructions self-reported in a pre-procedure questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kang X, Zhao L, Leung F, Luo H, Wang L, Wu J, Guo X, Wang X, Zhang L, Hui N, Tao Q, Jia H, Liu Z, Chen Z, Liu J, Wu K, Fan D, Pan Y, Guo X. Delivery of Instructions via Mobile Social Media App Increases Quality of Bowel Preparation. Clin Gastroenterol Hepatol. 2016 Mar;14(3):429-435.e3. doi: 10.1016/j.cgh.2015.09.038. Epub 2015 Oct 20. PMID 26492848
- [Result] Lee YJ, Kim ES, Choi JH, Lee KI, Park KS, Cho KB, Jang BK, Chung WJ, Hwang JS. Impact of reinforced education by telephone and short message service on the quality of bowel preparation: a randomized controlled study. Endoscopy. 2015 Nov;47(11):1018-27. doi: 10.1055/s-0034-1392406. Epub 2015 Jul 16. PMID 26182387